CLINICAL TRIAL: NCT02562274
Title: Evaluation of Consumption Safety and Effect of Mulberry Leaves and Vietnamese Coriander Based Instant Polyherbal Porridge on Working Memory and Bone Formation Markers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jintanaporn Wattanathorn, Associate Professor Doctor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HE 571373
Record Dates: First submitted 2015-09-18; First posted 2015-09-29 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Menopause; Cognitive impairment; Working memory; Bone formation markers; Osteoporosis
MeSH Terms: conditions — Cognitive Dysfunction; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Placebo Comparator): Subjects are received the placebo product which has same color and smell look like the herbal porridge containing the combined extract of mulberry and Vietnamese coriander (MP) treatments once daily for 8 weeks
  Interventions: Dietary Supplement: Placebo
- MP 50 mg/day (Active Comparator): Subjects are received the herbal porridge containing the combined extract of mulberry and Vietnamese coriander (MP) 50 mg/day treatments once daily for 8 weeks
  Interventions: Dietary Supplement: MP 50 mg/day
- MP 1500 mg/day (Active Comparator): Subjects are received the herbal porridge containing the combined extract of mulberry and Vietnamese coriander (MP) 1500 mg/day treatments once daily for 8 weeks
  Interventions: Dietary Supplement: MP 1500 mg/day

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects are received placebo treatments once daily for 8 weeks
  Arms: Placebo group
Dietary Supplement: MP 50 mg/day — Subjects are received MP 50 mg/day treatments once daily for 8 weeks
  Arms: MP 50 mg/day
Dietary Supplement: MP 1500 mg/day — Subjects are received MP 1500 mg/day treatments once daily for 8 weeks
  Arms: MP 1500 mg/day

SUMMARY:
This study the investigators aimed to determine the effect of the herbal porridge containing the combined extract of mulberry and Vietnamese coriander (MP) on cognitive function and bone formation markers of menopausal women. Forty-five participants were randomly assigned to receive a placebo or MP (50, 1500 mg) treatments once daily for 8 weeks.

DETAILED DESCRIPTION:
At present, the novel cheap and effective intervention against menopause related symptoms such as memory impairment and osteoporosis is still required due to the increased breast cancer risk induced by hormone replacement therapy. Based on the role of oxidative stress on cognitive deficit in menopause and the synergistic effect of herbs in traditional folklore, the cognitive enhancing effects and anti-osteoporosis effects of the functional food containing the combined extract of herbs possessing antioxidant effect has gained attention. Therefore, we aimed to determine the effect of the herbal porridge containing the combined extract of mulberry and Vietnamese coriander (MP) on cognitive function and bone formation markers of menopausal women. Forty-five participants were randomly assigned to receive a placebo or MP (50, 1500 mg) treatments once daily for 8 weeks. The cognitive function and working memory were assessed via the auditory oddball paradigm of event-related potentials and computerized battery tests respectively prior to the intervention, 1 month, 2 month, and at delay 1 month. Bone formation markers including serum calcium, alkaline phosphatase, and osteocalcin were determine prior to the intervention and at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy perimenopausal and postmenopausal women (<5 years menstruation cessation) who live in Northeastern of Thailand.
* Aged between 45-60 years old
* All volunteers don't have serious physical illness such as diabetes, high blood pressure, heart disease, liver disease, kidney disease, lung disease, allergies and mental disorder.
* All volunteers don't get medicine or hormone or other medicines that affect the nervous system and bone during the trial and within three months before the start of the test.
* All volunteers don't smoking more than 10 pieces/ day
* All volunteers don't have alcohol addiction
* On the day of the study, all volunteers felt well and refrain from drinking tea, coffee or alcohol at least 12 hour.

Exclusion Criteria:

* Volunteers who have been diagnosed with one of the following; cardiovascular diseases, respiratory diseases, neuropsychological diseases, head injury, diabetes mellitus, liver disease, cancer, autoimmune disease, hematological disorder, and gout or high uric acid.
* Volunteers who exposed to pesticides during one week before the test.
* Volunteers who have been Hysterectomy and/or Oophorectomy
* Volunteers who use hormone or any drug that effect on Hypothalamic Pituitary Gonadal axis and nervous system.
* Volunteers who require supplements or any drug that effect on the nervous system by order of the doctor during trial.
* Alcohol addiction
* Smoking addiction (smoking more than 10 pieces/ day)
* Athlete or volunteers who have a regular exercise more than 3 time/weeks
* Volunteers who don't follow instructions during the trial.
* Volunteers who participate in other projects.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Attention (N100) and cognitive processing (P300) determine by using Event Related Potential (Auditory oddball paradigm). | 3 months

SECONDARY OUTCOMES:
Accuracy and time response of working memory by using computerized batteries test (CDR) | 3 months
Bone formation marker by using serum calcium, serum alkaline phosphatase and serum osteocalcin | 2 months
Acetylcholinesterase and monoamine oxidase type A ,B activities in serum | 2 months
Psychological symptom by using SCL-90 questionnaire | 3 months
Consumption safety of MP product by using the electrocardiogram (ECG), hematology, blood chemistry and blood pressure measurement. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jintanaporn Wattanathorn, Ph.D., Principal Investigator — Khon Kaen University
Locations (1):
- Jitanaporn Wattanathorn, Khon Kaen, Changwat Khon Kaen, Thailand